#### INFORMED CONSENT TO PARTICIPATE IN RESEARCH

Please read the following information carefully. If you feel something is incorrect or unclear, please don't hesitate to ask for more information. If you agree with the proposal made to you, please sign this document.

#### 1. Research Title

Effectiveness of the INSIGHT Program: Intervention Program for those convicted of sexual crimes against children.

#### 2. Framework

This study takes place at the School of Psychology of the University of Minho within the scope of the Doctorate in Applied Psychology of Therapist Marta Sousa.

# 3. Study conditions

The program begins with a psychological assessment. Afterward, cases are randomly assigned to different working conditions. If you're in the intervention group, you immediately benefit from the program. If assigned to the control group, you can undertake the intervention if it demonstrates effectiveness.

The available intervention program is based on existing national and international literature, and is implemented over 25 sessions, in an individual format, on a weekly basis and lasting 60 minutes per session. Participation in this project is voluntary, subject to compliance with the following principles:

- 1) Completing a set of questionnaires, at the beginning, and at the end of the therapeutic process;
- 2) Completing a set of questionnaires three months after completing the intervention;
- 3) Compliance with weekly attendance (two consecutive absences will result in the completion of the process);
- 4) Carrying out Therapeutic Tasks between sessions.

Considering the voluntary nature of your participation, you may withdraw at any time without any consequences for you. Please note that you can be contacted, at the end of the intervention program, to carry out an interview about the therapeutic process.

## 4. CONDITIONS AND FINANCING

By participating in this study you will be contributing to the improvement of services provided in the context of this problem (deviant sexual behavior). Additionally, it will contribute to the carrying out of scientific studies within the scope of the Doctorate in Applied Psychology of Therapist Marta Sousa. No potential risks to your physical and/or psychological well-being are anticipated.

# 5. CONFIDENTIALITY AND ANONYMITY

All information collected will be treated confidentially. Only researchers involved in this project, with the consent of those responsible, will have access to the data.

| or any characteristic that could directly identify you will not be revealed. Furthermore, all data will be encoded using an identification number, which will allow other researchers accessing the data to only have access to that number, as well as generic sociodemographic data (e.g. age, profession). |
|---|
| Additional questions you may wish to ask after completing your participation can be asked to therapist Marta Sousa (e-mail: id9319@alunos.uminho.pt). |
| <u>Signature</u> : |
| I declare that I have read and understood this document, as well as the verbal information provided to me by the person signing above. I was guaranteed the possibility of, at any time, refusing to participate in this study without any consequences. Therefore, I agree to participate in this study and allow the use of the data that I voluntarily provide, trusting that they will only be used for this investigation and in the guarantees of confidentiality and anonymity given to me by the researcher. |
| Name: Signature: / / |
| I agree to the possibility of being contacted after the program to conduct a brief interview about my experience in the therapeutic process. |

When publishing works of a scientific nature, your identity will be protected, your name

THIS DOCUMENT IS COMPOSED OF TWO PAGES AND MADE IN DUPLICATE:

ONE WAY FOR THE INVESTIGATOR, ANOTHER WAY FOR THE CONSENTING PERSON